CLINICAL TRIAL: NCT05183984
Title: Randomized Study of Paclitaxel-carboplatin Followed by Niraparib Compared to Paclitaxel-carboplatin-bevacizumab Followed by Niraparib+bevacizumab in Patients with Advanced Ovarian Cancer, Following a Front-line Complete Surgery
Brief Title: Niraparib with BeVAcizumab After Complete CytoreductioN in Patients with OvArian Cancer
Acronym: NIRVANA-1
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GINECO-OV129b
Record Dates: First submitted 2021-11-22; First posted 2022-01-11 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; frontline surgery; brca status; maintenance
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Drug Therapy; Bevacizumab; niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A: carboplatin/paclitaxel + niraparib (Experimental): carboplatin AUC 5-6 + paclitaxel 175 mg/m² q3w, 5 cycles, followed by niraparib 200* or 300 mg/d for 2 years.
  Interventions: Drug: Chemotherapy; Drug: Niraparib
- ARM B: carboplatin/paclitaxel/bevaziumab + niraparib/bevacizumab (Experimental): carboplatin AUC 5-6 + paclitaxel 175 mg/m² + bevacizumab 15 mg/kg q3w, 5 cycles, followed by bevacizumab 15 mg/kg q3w for 15 months + niraparib 200*or 300 mg/d for 2 years.
  Interventions: Drug: Chemotherapy; Drug: Bevacizumab-Awwb; Drug: Niraparib

INTERVENTIONS:
Drug: Chemotherapy — Chemotherapy (carboplatin + paclitaxel) will be administred by intravenous infusion, AUC 5-6 q3w - 5 cycles during the treatment period
Drug: Bevacizumab-Awwb — MVASI (bevacizumab biosimilar) will be administrated by intravenous infusion at the second chemotherapy cycle for 5 cycles.
  the administration will continue during maintenance phase. Total bevacizumab duration therapy is 15 months.
  Arms: ARM B: carboplatin/paclitaxel/bevaziumab + niraparib/bevacizumab
Drug: Niraparib — niraparib will be administered orally once daily continuously after chemotherapy (+/- bevacizumab) cycles (maintenance treatment period). Total niraparib duration mainance treatment period is 2 years.

SUMMARY:
Randomized, open label, phase II multicenter study to assess the efficacy niraparib versus niraparib +bevacizumab maintenance in patients with newly diagnosed stage IIIA/B/C high-grade epithelial ovarian cancer with no residual disease after frontline surgery and treatment by adjuvant platinum-basedchemotherapy +/-bevacizumab.

DETAILED DESCRIPTION:
Phase II, randomized, open label, multicenterstudy.

Randomization on a 1:1 ratio, stratification performed according to:

BRCA status (local assessment) FIGO stage at diagnosis (IIIA versus IIIB/IIIC) Previous hyperthermic intraperitoneal chemotherapy (yes/no).

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patient should fulfill the following criteria:

1. Female patient ≥ 18 years of age.
2. Signed informed consent and ability to comply with treatment and follow-up.
3. Patient with newly diagnosed, a. Ovarian cancer, primary peritoneal cancer and/or fallopian-tube cancer, b. Histologically confirmed (based on local histopathological findings):

   • high grade serous or
   * high grade endometrioid (grade 2 and 3) or
   * other epithelial non mucinous and non-clear cell ovarian cancer in a patient with germline BRCA 1 or 2 deleterious mutation, c. At an advanced stage: FIGO stage IIIA to IIIC of the 2018 FIGO classification.
4. Patient having undergone frontline, complete cytoreductive surgery (i.e. no visible residual disease): The patient will be considered eligible once the ESGO Quality Assurance in Ovarian Cancer Surgery will have been filled out and validated
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. Patient must have received one cycle of carboplatin AUC 5-6 + paclitaxel 175 mg/m²
7. Patient must have started cycle 1 chemotherapy no later than 6 weeks after surgery.
8. Patient must have a thorax-abdomen-pelvis CT scan between surgery and Cycle 1, with no evidence of disease.
9. Patient eligible for first line platinum-taxane chemotherapy:
10. Patient eligible for bevacizumab treatment in combination with chemotherapy and in maintenance. It must be started at the second chemotherapy cycle and be administered at a dose of 15mg/kg every 3 weeks up to a total of 15 months.
11. Patient must have normal organ and bone marrow function before first cycle of chemotherapy:

    * Hemoglobin ≥ 9.0 g/dL.
    * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L.
    * Platelet count ≥ 100 x 109/L.
    * Total bilirubin ≤ 1.5 x institutional upper limit of normal (ULN).
    * Aspartate aminotransferase/Serum Glutamic Oxaloacetic Transaminase (ASAT/SGOT)) and Alanine aminotransferase /Serum Glutamic Pyruvate Transaminase (ALAT/SGPT)) ≤ 2.5 x ULN.
    * Serum creatinine ≤ 1. 5 x institutional ULN and GFR > 50 mL/min, by using an exact measure (ie. Iohexol clearance) or the most appropriate formula (Jeliffe, Cockroft Gault, MDRD, CKD-EPI) to the investigator's discretion.
    * Patient not receiving anticoagulant medication who has an International Normalized Ratio (INR) ≥1.5 and an Activated ProThrombin Time (aPTT) ≥1.5 x ULN.

    The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or APTT is within therapeutic limits (according to site medical standard). If the patient is on oral anticoagulants, dose has to be stable for at least two weeks at the time of randomization.
12. Urine dipstick for proteinuria < 2+. If urine dipstick is ≥2+, 24-hour proteinuria must be <1 g.
13. Normal blood pressure or adequately treated and controlled hypertension (systolic BP ≤ 140 mmHg and/or diastolic BP ≤ 90 mmHg).
14. Formalin fixed paraffin embedded (FFPE) tumor sample from the primary cancer must be available for local BRCA testing and if possible HRD testing (optional).
15. For countries where this will apply to: a subject will be eligible for randomization in this study only if either affiliated to, or a beneficiary of a social security category.

Exclusion Criteria:

* 1. Patient with clear cell adenocarcinoma or carcinosarcoma, non-epithelial origin of the ovarian tumor, the fallopian tube or the peritoneal tumor (i.e. germ cell tumors).

  2. Ovarian tumor of low malignant potential (e.g. borderline tumor), or mucinous carcinoma.

  3. Patient with a diagnosis, detection, or treatment of another type of cancer ≤ 3 years prior to initiating protocol therapy (except basal or squamous cell carcinoma of the skin and cervical cancer in situ that has been definitively treated and synchronous grade 1 stage 1 endometrial cancer) Patient with history of primary triple negative breast cancer may be eligible provided she completed her definitive anticancer treatment more than 3 years ago and she remains breast cancer disease free prior to start of study treatment.

  4. Patient with synchronous high grade serous or clear cell adenocarcinoma or carcinosarcoma of the endometrium is not eligible.

  5. Patient with myelodysplastic syndrome/acute myeloid leukemia history. 6. Patient receiving radiotherapy within 6 weeks prior to study treatment. 7. Previous allogenic bone marrow transplant. 8. Any previous treatment with PARP inhibitor. 9. Administration of other simultaneous chemotherapy drugs - except during a HIPEC procedure with cisplatin at PDS, any other anticancer therapy or anti-neoplastic hormonal therapy, or simultaneous radiotherapy during the trial treatment period (hormonal replacement therapy is permitted as are steroid antiemetics).

  10. Current or recent (within 10 days prior to randomization) chronic use of aspirin > 325 mg/day.

  11. Prior history of hypertensive crisis (CTC-AE grade 4) or hypertensive encephalopathy.

  12. Clinically significant (e.g. active) cardiovascular disease, including:
  * Myocardial infarction or unstable angina within ≤ 6 months of randomization,
  * New York Heart Association (NYHA) ≥ grade 2 congestive heart failure (CHF),
  * Poorly controlled cardiac arrhythmia despite medication (patient with rate controlled atrial fibrillation are eligible), or any clinically significant abnormal finding on resting ECG.
  * Peripheral vascular disease grade ≥ 3 (e.g. symptomatic and interfering with activities of daily living [ADL] requiring repair or revision).

    13. Previous Cerebro-Vascular Accident (CVA), Transient Ischemic Attack (TIA), Sub- Arachnoids Hemorrhage (SAH) or Posterior Reversible Encephalopathy Syndrome (PRES).

    14. History or evidence of hemorrhagic disorders. 15. Evidence of bleeding diathesis or significant coagulopathy (in the absence of coagulation).

    16. History or clinical suspicion of brain metastases or spinal cord compression. CT/MRI of the brain is mandatory (within 4 weeks prior to randomization) in case of suspected brain metastases. Spinal MRI is mandatory (within 4 weeks prior to randomization) in case of suspected spinal cord compression.

    17. History or evidence upon neurological examination of central nervous system (CNS) disease, unless adequately treated with standard medical therapy (e.g. uncontrolled seizures).

    18. Significant traumatic injury during 4 weeks prior to randomization. 19. Non-healing wound, active ulcer, or bone fracture. Patient with granulating incisions healing by secondary intention with no evidence of facial dehiscence or infection is eligible but require 3 weekly wound examinations.

    20. History of VEGF therapy related abdominal fistula or gastrointestinal perforation or active gastrointestinal bleeding within 6 months prior to the first study treatment.

    21. Current, clinically relevant bowel obstruction, including sub-occlusive disease, related to underlying disease.

    22. Patient with evidence of abdominal free air not explained by paracentesis or recent surgical procedure.

    23. Evidence of any other disease, metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment related complications.

    24. Pregnant or lactating women. 25. Participation in another clinical study with any intravenous or oral investigational product is not allowed. However, participation in a surgical clinical study including Hyperthermic Chemotherapy (HIPEC) during the surgical procedure is allowed.

    26. Patient unable to swallow orally administered medication and patient with gastrointestinal disorders likely to interfere with absorption of the study medication.

    27. Patient with a known contraindication or uncontrolled hypersensitivity to the components of paclitaxel, carboplatin, niraparib, bevacizumab, or their excipients.

    28. Immunocompromised patient, e.g., with known active hepatitis (i.e. Hepatitis B or C) due to risk of transmitting the infection through blood or other body fluids or patient who is known to be serologically positive for human immunodeficiency virus (HIV).

    29. Participant has a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2030-02 (Estimated)

PRIMARY OUTCOMES:
Progression-Free survival (PFS) rate up to 24 months | Progression-Free Survival (PFS) is defined as time from randomization until objective tumor progression or death, whichever occurs first, assessed up to 24 months.

SECONDARY OUTCOMES:
PFS2 | PFS2 is defined as time from randomization to objective tumor progression on next-line treatment or death from any cause, assessed up to 5 years.
Number of Participants with abnormal physical examinations, abnormal vital signs and abnormal findings according to CTC-AE v5 | Through treatment completion for all participants, an average of 28 months
Time to First Subsequent Treatment | TFST is defined as the time from the date of randomization to date of the first subsequent anticancer therapy or death, assessed up to 5 years.
Time to Second Subsequent Treatment | TSST is defined as the time from the date of randomization to the earlier of the date of second subsequent chemotherapy start date, or death date, assessed up to 5 years.
Long-term Overall Survival in both arms | from time of signature of informed consent, throughout the study period, assessed up to 5 years
Confirmation of the predictive value (overall chemo-sensitivity) of the KELIM. | From study start until the end of the study, assessed up to 5 years
  Repeated CA-125 assay repeated through study completion

CONTACTS AND LOCATIONS:
Overall Officials: Gilles FREYER, Pr, Principal Investigator — HCL - Centre Hospitalier Lyon Sud
Locations (87):
- France (49):
  - ICO Paul Papin, Angers
  - Sainte Catherine Institut du cancer Avignon-Provence, Avignon
  - CHRU Besançon - Hôpital Jean Minjoz, Besançon
  - Clinique Tivoli-Ducos, Bordeaux
  - Institut Bergonié, Bordeaux
  - Hôpital Morvan CHRU de Brest, Brest
  - HCL - Groupe Hospitalier Est, Bron
  - Centre François Baclesse, Caen
  - Centre Hospitalier de Cholet, Cholet
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU de Dijon - Bourgogne, Dijon
  - Centre Georges François Leclerc, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble - Institut Daniel Hollard, Grenoble
  - CHU Grenoble-Alpes - Site Nord (La Tronche), La Tronche
  - Clinique Victor Hugo, Le Mans
  - Centre Oscar Lambret, Lille
  - CHU de Limoges - Hôpital Dupuytren, Limoges
  - Centre Léon Bérard, Lyon
  - Hôpital Privé Jean Mermoz, Lyon
  - HCL - Hôpital de la Croix Rousse, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hôpital Nord Marseille, Marseille
  - Institut régional du cancer de Montpellier, Montpellier
  - CHU Montpellier - Hôpital Saint Eloi, Montpellier
  - Centre Azuréen de Cancérologie, Mougins
  - ORACLE - Centre d'Oncologie de Gentilly, Nancy
  - Hôpital Privé du Confluent, Nantes
  - Centre ONCOGARD - Institut de cancérologie du Gard, Nîmes
  - CHR Orléans, Orléans
  - Groupe Hospitalier Pitié Salpêtrière, Paris
  - Hôpital cochin, Paris
  - Hôpital Saint-Joseph, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Groupe Hospitalier Diaconesses - Croix Saint-Simon, Paris
  - Hôpital Tenon, Paris
  - HCL - Centre Hospitalier Lyon Sud (Hospices Civils de Lyon), Pierre-Bénite
  - Centre CARIO - HPCA, Plérin
  - CHU de Poitiers - Hôpital de la Milétrie, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - ICO - Centre René Gauducheau, Saint-Herblain
  - CHU de Saint-Etienne - Pôle de Cancérologie, Saint-Priest-en-Jarez
  - ICANS - Institut de cancérologie Strasbourg Europe, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - CHU Tours - Hôpital Bretonneau, Tours
  - CH Valence, Valence
  - Gustave Roussy, Villejuif
- Italy (5):
  - Firenze-Careggi, Florence
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Istituto Europeo di Oncologia (IEO), Milan
  - Ospedale San Gerardo Monza, Monza
  - Presidio Ospedaliero di Sondrio, Sondrio
- Japan (10):
  - Cancer Institute Hospital Of JFCR, Tokyo, Ariake, Koto
  - National Cancer Center Hospital East, Kashiwanoha, Chiba
  - Kurume University Hospital Clinical Research Center, Kurume, Fukuoka
  - University of Tsukuba Hospital, Tsukuba, Ibaraki-Pref
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Okayama University Hospital, Kita-ku, Okayama-ken
  - Jichi Medical UH, Shimotsuke, Tochigi
  - Ehime University Hospital, Ehime, Toonshi
  - Yamagata University Hospital, Yamagata, Yamagata
  - Saitama Medical University International Medical Center, Saitama
- Singapore (2):
  - National University Hospital (NUH), Singapore
  - National Cancer Centre Singapore, Singapore
- South Korea (5):
  - Samsung Medical Center, Seoul, Gangnam-gu
  - National Cancer Center, Seoul, Gyeonggi-do
  - National University Hospital, Seoul, Jongno-gu
  - Severance Hospital, Seoul, Seodaemun-gu
  - Asan Medical Center, Seoul, Songpa-gu
- Spain (16):
  - Coruña University Hospital (CHUAC), A Coruña
  - Hospital del Mar, Barcelona
  - Hospital Universitari Dexeus, Barcelona
  - Hospital San Pedro de Alcantara, Cáceres
  - Hospital Clínico Universitario Virgen de la Arrixaca, El Palmar, Murcia
  - Hospital Universitario de Jerez, Jerez de la Frontera
  - Clínica Universidad de Navarra, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Virgen de la Victoria, Málaga
  - Hospital Universitario Central de Asturias, Oviedo
  - Clinica Universidad de Navarra., Pamplona
  - Complejo Hospitalario de Navarra, Pamplona
  - CHU de Santiago de Compostela, Santiago de Compostela
  - Hospital Universitari MutuaTerrassa, Terrassa
  - Fundación Investigación Clínico de Valencia., Valencia

REFERENCES:
- [Derived] Sghaier S, Corbaux P, Ray-Coquard I, Lim MC, Hasegawa K, Nieuwenhuysen EV, Gonzalez A, Raspagliesi F, Freyer G. NIRVANA-1: maintenance therapy with niraparib versus niraparib-bevacizumab in patients with advanced ovarian cancer. Future Oncol. 2023 Aug;19(25):1715-1727. doi: 10.2217/fon-2023-0167. Epub 2023 Aug 31. PMID 37650734